CLINICAL TRIAL: NCT02409108
Title: An Early Feasibility Study of Perfusion-Induced Hyperthermia for Metastatic Non-Small Cell Lung Carcinoma and All Relapsed Malignancies, for Which Curative Therapy is Not Possible
Brief Title: Perfusion-Induced Hyperthermia for Metastatic Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Kiev (Other)
Collaborators: Exatherm, Inc (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Kiev, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MCC-14-0929-F3R; 2014-089 (Other: University of Kentucky)
Record Dates: First submitted 2015-03-17; First posted 2015-04-06 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Non-Small Cell Lung Carcinoma; Solid Tumor, Adult
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Exatherm-TBH system (Experimental): One treatment of Total Body Hyperthermia
  Interventions: Device: Exatherm-TBH system

INTERVENTIONS:
Device: Exatherm-TBH system — One treatment of Total Body Hyperthermia

SUMMARY:
The purpose of this study is to gather information on how safe the hyperthermia treatment delivered via the Exatherm-TBH (the device that will heat your blood and deliver it back to you), added to the best supportive care is to patients who have advanced persistent or recurrent, unresectable Cancer.

DETAILED DESCRIPTION:
One potential candidate for a new approach to advanced cancer therapy is hyperthermia because cancer cells are thermo-sensitive, with significantly reduced heat shock protein (HSP) expression. Moreover, hyperthermia (42°C) causes repression of genes involved in the cell cycle and cellular growth and proliferation. Upon exposure to hyperthermic conditions, HSP expression is increased in normal cells. However, when cancer cells are exposed to hyperthermia, they initially express significantly less HSPs than normal cells, which sensitizes them to hyperthermia. Mild hyperthermia (43°C for less than two hours) induces extensive double-stranded DNA fragmentation and, at a later time, apoptosis in murine thymocytes. In cells with irreparable levels of DNA damage, apoptosis is the means of elimination.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of Stage IIIB or Stage IV of non-small cell lung cancer and have received at least two lines of FDA-approved or National Comprehensive Cancer Network (NCCN) accepted systemic therapy and progressed through, or not tolerated, such therapy.

  * Subjects whose tumors harbor an exon 19 deletion or exon 21L858R EGFR mutation must have progressed on or had intolerance to EGFR tyrosine kinase inhibitor.
  * Subjects whose tumors harbor an AKL translocation must have progressed on or had intolerance to crizotinib (or any FDA approved ALK inhibitor).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2

  * Have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective

Must have undergone at least 2 prior regimens for treatment of recurrent or metastatic disease

* Life expectancy of greater than 3 months.
* Age ≥22 years.
* There is no restriction on the number of prior therapies allowed for this disease and prior radiation and chemotherapy is allowed, provided the subject has recovered from all grade 2 or greater toxicity prior to enrollment.
* Patient understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provide written informed consent prior to the procedure

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C, or monoclonal antibodies such as bevacizumab, cetuximab or panitumumab) prior to entering the study or those who have not recovered to < grade 2 adverse events due to agents administered more than 4 weeks earlier.
* Patients with stroke or TIA within 90 days prior to enrollment; or peripheral vascular disease requiring intervention within the 90 days prior to enrollment; or any known hemodynamically significant lesion or embolic plaque.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * total Bilirubin, AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * glomerular filtration rate (GFR)> 60 as defined by the Modification of Diet in Renal Disease (MDRD) formula
  * Thromboplastin Time (PTT) < 35 sec)
* Patients with uncontrolled seizure disorder, spinal cord compression or carcinomatous meningitis.
* Patients with a mental disorder, psychiatric illness/social or concussion which would inhibit their ability to provide informed consent or prevent compliance with follow-up.
* Patients with high risk of cardiovascular event such as severe uncontrolled hypertension (>170/110 systemic blood pressure on therapy), or pulmonary hypertension (greater than .5 systolic blood pressure
* ST elevation myocardial infarction within 30 days prior to enrollment; unstable angina or significant, untreated arrhythmias within 30 days prior to enrollment.
* Patients with moderate to severe heart failure, New York Heart Association (NYHA) class III or IV, liver dysfunction with total bilirubin >2. 5 upper limit of normal, or serum creatinine >2.5 mg/dL or any form of dialysis; within 30 days prior to enrollment.
* Patients with a major surgical procedure or other investigational agents within 30 days before study enrollment.
* Patients with known, untreated or progressive brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Pregnant women are excluded from this study
* Patients with documented contraindication to anticoagulation therapy such as heparin induced thrombocytopenia or a documented coagulopathy or hematologic disorder that would contraindicated undergoing treatment and use of the associated anticoagulant agents required during treatment.
* Patients with documented active bacterial, viral or fungal infection, untreated systematic peptic ulcer disease, uncontrolled diabetes mellitus or serious concurrent medical disease that could limit survival to less than 3 months.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for harm when exposed to hyperthermia, as well as negative interactions of these medications with hyperthermia.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-02-16 (Actual)

PRIMARY OUTCOMES:
Safety as measured by adverse events | Up to 12 weeks after treatment
  Incidence of adverse events as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4.0. Adverse event data and corresponding toxicity grades during treatment will be summarized in the form of tables. Incidence tables will be generated to summarize incidence of patients reporting at least one episode of each specific adverse event, incidence of adverse events causing withdrawal and incidence of serious adverse event. The total number of episodes for each event reported (Frequency Table), the severity and attribution to study therapy of each episode reported (Severity Table and Attribution Table) will also be displayed. Safety data will be summarized for the overall treated group and the overall concurrent control group. Reversibility of the adverse events and toxicities will also be summarized.
Exatherm-TBH device functionality | Time frame: day 1
  Device functionality will be documented and summarized using descriptive statistics and presented in the form of tables
Safety as measured by serious adverse events | Up to 12 weeks after treatment
  Incidence of serious adverse events associated with hyperthermic treatment as graded by the NCI CTCAE v. 4.0. Summarized in the form of tables. Listings of adverse events by patients will include the time to onset, the duration of each event, the severity of each event, and the relationship of the event to study therapy, whether it was a serious event, and whether it caused withdrawal.
Quality of Life | Baseline and up to 1 year after treatment
  Assess changes in quality of life as documented by the EQ-DL-3L. QOL and neurocognitive testing will be summarized using descriptive statistics including mean, median and variation levels of QOL score
Complication rates associated with hyperthermic treatment | Up to 12 weeks post-treatment
  Complication rates will be documented and summarized using descriptive statistics and presented in the form of tables

SECONDARY OUTCOMES:
Response rate | Up to 12 weeks after treatment
  Assess clinical benefit rate as documented by CR+PR+SD.
Time to treatment failure | Up to 12 weeks after treatment
  Documentation of disease progression presented with Kaplan Meier curve.
Progression free survival | Baseline up to 1 year
  Progression free survival following hyperthermic therapy presented with Kaplan Meier curve
Death | Baseline up to 1 year
  Documentation of time of death presented with Kaplan Meier curve

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kiev, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky, Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No